CLINICAL TRIAL: NCT07291544
Title: Management of Supraventricular Tachycardias in Children: A National Multicenter Study
Brief Title: Management of Supraventricular Tachycardias in Children
Status: Completed | Type: Observational
Sponsor: Paris Cardiovascular Research Center (Inserm U970) (Other Government)
Responsible Party: Principal Investigator, Victor WALDMANN, Head of pediatric and congenital electrophysiology, Paris Cardiovascular Research Center (Inserm U970)
Other Study IDs: WALDMANN202501
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Supraventricular Arrhythmias; Children; Management
Keywords: supraventricular arrhythmias; supraventricular tachycardia; children
MeSH Terms: conditions — Tachycardia, Supraventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Management of children with supraventricular tachycardias — Observational analysis of the management of supraventricular tachycardias (antiarrhythmic drugs and catheter ablations)

SUMMARY:
Background

Supraventricular tachycardias (SVTs) are the most common arrhythmic events in children, with an estimated incidence of 13 per 100,000 per year before the age of 18. Few large patient cohorts have been reported, as most published studies are single-center. Large-scale studies come from medico-administrative databases, which lack the granularity needed for detailed analysis of outcomes according to the therapies used and the type of SVT.

Furthermore, although a large proportion of neonatal SVTs do not recur (spontaneous resolution of the accessory pathway), there are limited comparative data on the effectiveness of antiarrhythmic therapies specifically in children after the age of 1 year. Management therefore varies greatly, in part because current guidelines propose different therapeutic options based on low-level evidence.

Objectives:

* Describe the management of SVTs (antiarrhythmic therapies and catheter ablation) in children in France
* Compare the effectiveness of different antiarrhythmic treatments according to age (<1 year and >1 year) and type of SVT
* Analyze the incidence of adverse events and complications associated with antiarrhythmic treatments and catheter ablation

ELIGIBILITY:
Inclusion Criteria:

* Age <18 years at the time of the first documented supraventricular tachycardia episode

Exclusion Criteria:

* Early postoperative supraventricular tachycardia (<30 days)
* Age ≥18 years at the first documented supraventricular tachycardia episode
* Fetal tachycardias without postnatal recurrence
* Atrial extrasystoles without sustained runs (<30 seconds)

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children <18 years old with a documented episode (ECG, Holter-ECG, wearable device, or implantable device) of sustained SVT (>30 seconds) will be eligible. Although most children in this context do not have structural heart disease, those with congenital or structural heart disease will also be eligible. Participation will be proposed to all pediatric cardiology centers in France through the Filiale de Cardiologie Pédiatrique et Congénitale (FCPC).
Sampling Method: Probability Sample
Enrollment: 1400 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Antiarrhythmic therapies | At the time of the first supraventricular tachycardia recorded
  Proportion of antiarrhythmic therapies used by age group (<1 year and >1 year)
Catheter ablation | At the time of first episode of supraventricular tachycardia or after recurrence
  Proportion of children referred for catheter ablation and age at ablation
Recurrence of supraventricular tachycardia | At 1 year after antiarrhythmic drug initiation
  Time between antiarrhythmic therapy initiation and first recurrence, according to treatment and age

IPD SHARING:
Plan to Share IPD: No